CLINICAL TRIAL: NCT05325281
Title: A Phase I Dose-Escalation Study of CPI-613 (Devimistat) in Combination With Chemoradiation in Patients With Pancreatic Adenocarcinoma
Brief Title: CPI-613 (Devimistat) in Combination With Chemoradiation in Patients With Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmaceutical funder pulled funding and no longer plans to develop the drug further.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Cornerstone Pharmaceuticals (Industry); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Mandana Kamgar, MD, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00043904
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pancreas Adenocarcinoma
Keywords: CPI-613; Devimistat; intensity-modulated radiation therapy
MeSH Terms: interventions — devimistat; Gemcitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CPI-613® (Dose level -1.0 250 mg/m^2) (Experimental): Dose escalation/de-escalation for CPI-613® (devimistat) will be conducted using a Bayesian optimal interval (BOIN) design. Gemcitabine will be infused over 30 minutes at a fixed dose of 400 mg/m^2 weekly. Intensity-modulated radiation therapy will be administered at 54 Gy in 30 fractions of 1.8 Gy per fraction, with five fractions given per week. CPI-613® will be given once per week by IV infusion.
  Interventions: Drug: CPI-613® (Dose level -1.0 250 mg/m^2); Drug: Gemcitabine; Radiation: Intensity-modulated Radiation Therapy
- CPI-613® (Dose level 1.0 500 mg/m^2) (Experimental): Dose escalation/de-escalation for CPI-613® (devimistat) will be conducted using a Bayesian optimal interval (BOIN) design. Gemcitabine will be infused over 30 minutes at a fixed dose of 400 mg/m^2 weekly. Intensity-modulated radiation therapy will be administered at 54 Gy in 30 fractions of 1.8 Gy per fraction, with five fractions given per week. CPI-613® will be given once per week by IV infusion.
  Interventions: Drug: CPI-613® (Dose level 1.0 500 mg/m^2); Drug: Gemcitabine; Radiation: Intensity-modulated Radiation Therapy
- CPI-613® (Dose level 2.0 1,000 mg/m^2) (Experimental): Dose escalation/de-escalation for CPI-613® (devimistat) will be conducted using a Bayesian optimal interval (BOIN) design. Gemcitabine will be infused over 30 minutes at a fixed dose of 400 mg/m^2 weekly. Intensity-modulated radiation therapy will be administered at 54 Gy in 30 fractions of 1.8 Gy per fraction, with five fractions given per week. CPI-613® will be given once per week by IV infusion.
  Interventions: Drug: CPI-613® (Dose level 2.0 1,000 mg/m^2); Drug: Gemcitabine; Radiation: Intensity-modulated Radiation Therapy
- CPI-613® (Dose level 3.0 1,500 mg/m^2) (Experimental): Dose escalation/de-escalation for CPI-613® (devimistat) will be conducted using a Bayesian optimal interval (BOIN) design. Gemcitabine will be infused over 30 minutes at a fixed dose of 400 mg/m^2 weekly. Intensity-modulated radiation therapy will be administered at 54 Gy in 30 fractions of 1.8 Gy per fraction, with five fractions given per week. CPI-613® will be given once per week by IV infusion.
  Interventions: Drug: CPI-613® (Dose level 3.0 1,500 mg/m^2); Drug: Gemcitabine; Radiation: Intensity-modulated Radiation Therapy
- CPI-613® Maximum Tolerated Dose (MTD) (Experimental): MTD of CPI-613® from initiation of treatment to 30 days after treatment. MTD will be determined by testing increasing doses of CPI-613®, starting from 500 mg/m^2 and up to 1,500 mg/m^2, on dose escalation cohorts of three patients (maximum 24 patients) in combination with Gem-RT therapy. MTD reflects the highest drug dose that does not cause unacceptable adverse effects, with a target dose-limiting toxicity (DLT) rate of 30%. Final dose will be revised as appropriate.
  Interventions: Drug: CPI-613® (Dose level -1.0 250 mg/m^2); Drug: CPI-613® (Dose level 1.0 500 mg/m^2); Drug: CPI-613® (Dose level 2.0 1,000 mg/m^2); Drug: CPI-613® (Dose level 3.0 1,500 mg/m^2); Drug: CPI-613® Maximum Tolerated Dose (MTD); Drug: Gemcitabine; Radiation: Intensity-modulated Radiation Therapy

INTERVENTIONS:
Drug: CPI-613® (Dose level -1.0 250 mg/m^2) — CPI-613® is a mitochondrial metabolism inhibitor. CPI-613® is a lipoic acid antagonist that abrogates mitochondrial energy metabolism to induce apoptosis in various cancer cells.
  Other Names: Devimistat; alpha-lipoic acid analogue CPI-613
  Arms: CPI-613® (Dose level -1.0 250 mg/m^2); CPI-613® Maximum Tolerated Dose (MTD)
Drug: CPI-613® (Dose level 1.0 500 mg/m^2) — CPI-613® is a mitochondrial metabolism inhibitor. CPI-613® is a lipoic acid antagonist that abrogates mitochondrial energy metabolism to induce apoptosis in various cancer cells.
  Other Names: Devimistat; alpha-lipoic acid analogue CPI-613
  Arms: CPI-613® (Dose level 1.0 500 mg/m^2); CPI-613® Maximum Tolerated Dose (MTD)
Drug: CPI-613® (Dose level 2.0 1,000 mg/m^2) — CPI-613® is a mitochondrial metabolism inhibitor. CPI-613® is a lipoic acid antagonist that abrogates mitochondrial energy metabolism to induce apoptosis in various cancer cells.
  Other Names: Devimistat; alpha-lipoic acid analogue CPI-613
  Arms: CPI-613® (Dose level 2.0 1,000 mg/m^2); CPI-613® Maximum Tolerated Dose (MTD)
Drug: CPI-613® (Dose level 3.0 1,500 mg/m^2) — CPI-613® is a mitochondrial metabolism inhibitor. CPI-613® is a lipoic acid antagonist that abrogates mitochondrial energy metabolism to induce apoptosis in various cancer cells.
  Other Names: Devimistat; alpha-lipoic acid analogue CPI-613
  Arms: CPI-613® (Dose level 3.0 1,500 mg/m^2); CPI-613® Maximum Tolerated Dose (MTD)
Drug: CPI-613® Maximum Tolerated Dose (MTD) — MTD will be determined by testing increasing doses of CPI-613®, starting from 500 mg/m^2 and up to 1,500 mg/m^2, on dose escalation cohorts of three patients (maximum 24 patients) in combination with Gem-RT therapy. MTD reflects the highest drug dose that does not cause unacceptable adverse effects, with a target dose-limiting toxicity (DLT) rate of 30%. Final dose will be revised as appropriate.
  Other Names: Devimistat; alpha-lipoic acid analogue CPI-613
  Arms: CPI-613® Maximum Tolerated Dose (MTD)
Drug: Gemcitabine — Subjects will be administered 400 mg/m^2 gemcitabine once per week by IV infusion over approximately 30 minutes for six weeks.
  Other Names: Gemzar®
Radiation: Intensity-modulated Radiation Therapy — 1.8 Gy per fraction, 5 fractions per week, 30 fractions total (54 Gy) across six weeks.

SUMMARY:
This is a single-center, open-label, phase I study designed to determine the maximum tolerated dose (MTD) and safety profile of CPI-613® when used concomitantly with chemoradiation for local control of pancreatic adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
This study is designed to test the hypothesis that a combination of gemcitabine and radiation therapy (Gem-RT) with CPI-613®, a selective mitochondrial metabolism inhibitor in PDAC tumor cells, will be well tolerated without additional significant toxicity. Additionally, CPI-613® is expected to improve the Gem-RT effectiveness, resulting in durable local control of disease. As a necessary and initial step to translate preclinical observations into a patient setting and test our proposed hypotheses, the investigators will perform a dose-finding phase I clinical trial that has been designed to evaluate the maximum tolerated dose (MTD), recommended phase II dose (RP2D), and safety profile of CPI-613® along with standard of care Gem-RT in patients with unresectable PDAC in need of definitive local control of disease. The overarching goals for this trial are to determine the safety and toxicity of CPI-613® when given concurrently with Gem-RT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Pathologically confirmed (histologic or cytologic) adenocarcinoma of the pancreas.
3. Patients should have an inoperable disease (locally advanced, oligometastatic, or medically inoperable) and, based on the review of the institutional pancreatic tumor board, should otherwise benefit from chemoradiation for definitive local control of the primary tumor.
4. Patients with and without regional adenopathy are eligible.
5. History/physical examination, including a collection of weight and vital signs, within 30 days prior to treatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within 14 days of study entry.
7. Imaging requirements are to include

   1. Diagnostic abdominal/pelvic CT with IV contrast or abdominopelvic magnetic resonance (MR) scan with perfusion and diffusion-weighted sequences within 45 days prior to study entry.
   2. Chest CT scan or X-ray within 45 days prior to study entry.
   3. Radiation treatment planning abdominal CT. A recommended abdominal MR will be done as a simulation (SIM) scan with interpretation. The CT SIM will not be done with interpretation. Positron emission tomography (PET) scan and MRI are both optional but encouraged. Abdominal MR scans for staging and radiation planning and follow-up are optional but encouraged.
8. Heme Onc (Chem 24) and cancer antigen 19-9/ carcinoembryonic antigen (CEA) within 30 days prior to treatment, as follows:

   1. Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3.
   2. Platelets ≥ 100,000 cells/mm3.
   3. Hemoglobin ≥ 8.0g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin ≥ 8.0 g/dl is acceptable).
   4. Not on hemodialysis.
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <4x the upper limit of normal.
   6. Total bilirubin <2x the upper normal mg/dL (higher levels are acceptable if Gilbert Syndrome is suspected clinically).
9. Negative serum pregnancy test (if applicable).
10. Ability to position for radiation therapy.
11. Pregnancy It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female patients participating in this study should avoid becoming pregnant, and male patients should avoid impregnating a female partner. Non-sterilized female patients of reproductive age and male patients should use effective methods of contraception through defined periods during and after study treatment as specified below.

    Female patients must meet one of the following:
    * Postmenopausal for at least one year before the screening visit, or
    * Surgically sterile, or
    * If they are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through three months after the last dose of study drug, and
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)

    Male patients, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:
    * Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, or
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
12. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Prior invasive malignancy (except nonmelanomatous skin cancer, noninvasive breast cancer [ductal carcinoma in situ], or prostate cancer under active surveillance). Other malignancies are allowed if the patient has been disease free for a minimum of two years.
2. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
3. Any major surgery within 28 days prior to study entry, except colonic stent placement, intestinal diversion without resection, exploratory laparotomy and laparoscopy or vascular access insertion.
4. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during the course of the study and for women three months after study therapy is completed and for men six months after study therapy is completed. This exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
5. Life expectancy less than two months.
6. Severe, active co-morbidity, defined as follows:

   * Any unresolved bowel or bile duct obstruction, or
   * Symptomatic myocardial ischemia, or
   * uncontrolled clinically significant conduction abnormalities (e.g., ventricular tachycardia on antiarrhythmics is excluded and first-degree atrioventricular (AV) block or asymptomatic left anterior fascicular block (LAFB) / right bundle branch block (RBBB) will not be excluded), or
   * Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose
   * Any active uncontrolled bleeding or patients with a bleeding diathesis.
7. Serious psychiatric illness (e.g., depression, psychosis) or medical conditions that in the opinion of investigator could interfere with treatment.
8. Concurrent therapy with approved or investigational anticancer therapeutics other that what is stipulated by the protocol.
9. Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) RNA or HBsAg (HBV surface antigen).
10. Known to be HIV seropositive and on anti-HIV drugs because of the unknown interactions between these drugs and the study agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of CPI-613® | Initiation of treatment to 30 days after treatment
  MTD will be determined by testing increasing doses of CPI-613®, starting from 500 mg/m^2 and up to 1,500 mg/m^2, on dose escalation cohorts of three patients (maximum 24 patients) in combination with Gem-RT therapy. MTD reflects the highest drug dose that does not cause unacceptable adverse effects.

SECONDARY OUTCOMES:
The number of subjects with adverse events related to the treatment | Start of study treatment until 30 days after completion of study treatment.
  All adverse events will be documented using the NCI CTCAE version 5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Kamgar, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan HY, Kamgar M, Aboukameel A, Bannoura S, Chung BY, Li Y, Hallak MNA, Philip PA, Tsai S, Luther S, Hall WA, Azmi AS. Targeting Cellular Metabolism With CPI-613 Sensitizes Pancreatic Cancer Cells to Radiation Therapy. Adv Radiat Oncol. 2022 Nov 9;8(1):101122. doi: 10.1016/j.adro.2022.101122. eCollection 2023 Jan-Feb. PMID 36479231